CLINICAL TRIAL: NCT05087550
Title: Multicenter Study on Organ Acquisition Costs in the Post Re-Allocation Era: Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 058.HPB.2021.D
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-08

CONDITIONS: Liver Transplant
Keywords: Organ Procurement and Transplant Network (OPTN); Liver Allocation Policy
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver Transplantation patients
  Interventions: Procedure: Liver Transplantation

INTERVENTIONS:
Procedure: Liver Transplantation — Patients who underwent liver transplantation at Methodist Dallas Medical Center

SUMMARY:
Organ procurement organizations (OPO) have increased organ recovery efficiency and yield and have also reduced organ acquisition charges. The new liver allocation policy came into effect in February 2020 and aims to increase access to organs for waitlist candidates with the greatest severity of illness. The urgent change was driven by the perception that patients were dying because of arbitrary boundaries and inequitable access. Critics of the new policy have highlighted the potential cost implications particularly at an OPO level. A study of five OPOs throughout the United States highlighted an increase in costs ranging from 43% - 206% despite the same volume of livers transplanted. The main reason for the cost appears to lie in organ handling and transport. This mirrors the findings of Puri and colleagues who acknowledged changes to lung transplantation at Barnes Jewish Hospital in the pre- and post-policy eras and reported a substantial decline in local donors. The new lung system has also resulted in a higher organ discard rate and ultimately higher costs. Such data has generated meaningful discussions regarding optimizing organ allocation polices, however, data from individual transplant centers is lacking in the literature. Changes at a transplant center level relating to recipient costs are likely impacted by the new policy, which could be related to patient travel, accommodation, work up etc.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Underwent liver transplantation at MDMC between February 4th 2019 - February 4th 2020 and February 5th 2020 - February 5th 2021

Exclusion Criteria:

* Below 18 years of age
* Did not undergo liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from patients who underwent liver transplantation between February 4th, 2019 - February 4th, 2020, and February 5th, 2020 - February 5th, 2021 will be included in the study.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Liver transplant volume | 02/04/2019 - 02/05/2021
Cost | 02/04/2019 - 02/05/2021
  Costs related to:
  * Transplant volume and organ recovery information
  * Transportation costs, distance traveled, travel time
  * Personnel costs
  * Hospital charges/costs

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Mejia, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No